CLINICAL TRIAL: NCT05487768
Title: Functional Connectivity After Anterior Cruciate Ligament Reconstruction
Acronym: FCACLR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ONZ-2022-0231
Record Dates: First submitted 2022-07-27; First posted 2022-08-04 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Anterior Cruciate Ligament Rupture; Electroencephalography; Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anterior cruciate ligament reconstruction group (Experimental): Patients that underwent an anterior cruciate ligament reconstruction
  Interventions: Other: EEG measurement
- Control group (Active Comparator): Healthy matched controls
  Interventions: Other: EEG measurement

INTERVENTIONS:
Other: EEG measurement — EEG measurement to evaluate functional connectivity in the brain during 3 motor tasks:
  * Knee extension while sitting (10x left - right)
  * Bipodal squatting (10x)
  * Unipodal stance (5x30 seconds left-right)

SUMMARY:
Background:

Despite surgical reconstruction and rehabilitation, individuals after a primary anterior cruciate ligament injury have a significantly increased risk of relapse. The mechanisms for this increased risk may go beyond mere physiological and biomechanical changes of the reconstructed anterior cruciate ligament. The loss of ligamentous mechanoreceptors can affect sensory feedback and consequently result in a disrupted afferent input to the central nervous system. However, research on the neuroplasticity of the central nervous system after anterior cruciate ligament injury and more specifically on the cooperation between different brain areas (=functional connectivity) in motor execution and performance is limited.

Research purpose:

To investigate the changes in terms of functional connectivity in the brain after sustaining an anterior cruciate ligament injury and associated reconstruction?

Population:

* Patients after anterior cruciate ligament reconstruction
* Healthy controls

Protocol:

First, all participants are required to complete several questionnaires regarding the level of anxiety and the functioning of the knee in daily activities and sports. In addition, during the baseline testing, participants will be required to perform an experiment while electrical brain activity is recorded by means of an electroencephalography (EEG) measurement. During this experiment, the participants will have to successively perform the following exercises: 10x knee extension from sitting (left and right), 10x bipodal squat from standing, 5x 30 seconds unipodal standing (left and right).

The above protocol will be administered to the patient group for the first time 8 weeks after the anterior cruciate ligament reconstruction. When the patients do not need further rehabilitation, they will be invited a second time to execute the same protocol again. The control group will only have to carry out the above protocol once.

Finally, for one year after the last test, the patient group will be contacted monthly to monitor return to sport and the occurrence of injuries.

ELIGIBILITY:
PATIENT GROUP

Inclusion Criteria:

* Older than 18 years of age.
* Primary anterior cruciate ligament rupture and reconstruction

Exclusion Criteria:

* Major knee surgery in the past.
* Diagnosed with any knee pathology at this moment.
* Have any muscle or nerve related conditions that affect the functioning of the lower limbs.

CONTROL GROUP

Inclusion Criteria:

- Older than 18 years of age.

Exclusion Criteria:

* Major knee surgery in the past.
* Diagnosed with any knee pathology at this moment.
* Have any muscle or nerve related conditions that affect the functioning of the lower limbs.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change in functional connectivity in the brain in patients following anterior cruciate ligament reconstruction | Experimental group: 8 weeks postoperative and at the end of the rehabilitation (on average 9-12 months postoperative) / Control group: baseline
  Electroencephalography (EEG) will be recorded from a 128 Sn surface electrode cap during 3 motor tasks. Functional connectivity will be analyzed.

SECONDARY OUTCOMES:
Change in subjective knee functionality measured by the Knee injury and Osteoarthritis Outcome Score (KOOS) - Questionnaire | Experimental group: 8 weeks postoperative and at the end of the rehabilitation (on average 9-12 months postoperative) / Control group: baseline
  Assess the patients opinion about their knee and associated problems. Each item is given a score between 0 and 4, then the total score is converted to a scale of 0-100. A higher score indicates less disfunction.
Change in kinesiophobia measured by the Tampa scale of Kinesiophobia (TSK) - Questionnaire | Experimental group: 8 weeks postoperative and at the end of the rehabilitation (on average 9-12 months postoperative) / Control group: baseline
  This questionnaire consists of 17 questions and evaluates the extent to which patients experience kinesiophobia.
  Each item is given a score between 0 and 4. A higher score indicates more kinesiophobia.
Change in knee confidence - Questionnaire | Experimental group: 8 weeks postoperative and at the end of the rehabilitation (on average 9-12 months postoperative) / Control group: baseline
  To evaluate the confidence of patients in their operated knee, expressed as a percentage relative to the nonoperated side (0-100%). A lower score indicates less confidence.
Change in worrying behaviour measured by the Penn State Worry Questionnaire (PSWQ) - Questionnaire | Experimental group: 8 weeks postoperative and at the end of the rehabilitation (on average 9-12 months postoperative) / Control group: baseline
  This questionnaire consists of 16 questions and evaluates the extent to which patients are concerned
  Each item is given a score between 1 and 5. The total scores range from 16 to 80 with higher scores indicative of higher levels of trait worry.
Change in athletes' emotion, confidence, and risk appraisal when returning to sports after an anterior cruciate ligament reconstruction measured by the ACL-Return to sport after injury (ACL-RSI) - Questionnaire | Experimental group: 8 weeks postoperative and at the end of the rehabilitation (on average 9-12 months postoperative) / Control group: baseline
  This questionnaire consists of 12 questions divided into three main sections: athletes' emotion, confidence, and risk assessment when returning to sport after an ACL injury and/or reconstructive surgery.
  Each item is given a score between 0 and 100, after which the total score is converted to a scale of 0-100. A lower score indicates more concerns about return to sport.
Follow up questionnaire | Monthly, for one year after the end of the rehabilitation (on average 9-12 months postoperative).
  To monitor return to sport and injury occurence in the patient group

CONTACTS AND LOCATIONS:
Overall Officials: Erik Witvrouw, Prof. Dr., Principal Investigator — Department of Rehabilitation Sciences, Ghent University
Locations (1):
- Ghent University, Department of Rehabilitation Sciences, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No